CLINICAL TRIAL: NCT00509470
Title: ONgoing Evaluation of Depressor Effect And Safety of Combination Therapy With Telmisartan and Low-dose Hydrochlorothiazide in Patients With Hypertension Uncontrolled on Amlodipine Treatment
Brief Title: Evaluation of Effect of Combination With Telmisartan and Hydrochlorothiazide in Hypertensives Uncontrolled on Amlodipine
Acronym: ONEAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tokyo University (Other)
Responsible Party: Principal Investigator, Hiroshi Satonaka, Professor, Tokyo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2007008
Record Dates: First submitted 2007-07-28; First posted 2007-07-31 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Telmisartan; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- telmisartan plus low-dose hydrochlorothiazide (Active Comparator): 12 week combination therapy with telmisartan plus low-dose hydrochlorothiazide
  Interventions: Drug: telmisartan plus hydrochlorothiazide
- Amlodipine (Active Comparator): Amlodipine is continuously administered.
  Interventions: Device: Amlodipine

INTERVENTIONS:
Drug: telmisartan plus hydrochlorothiazide — Combination therapy with telmisartan (40 mg/day) plus hydrochlorothiazide (12.5 mg/day): If blood pressure is not reach to lower than 140/90 mmHg, dose of telmisartan can be increased to 80 mg/day
  Arms: telmisartan plus low-dose hydrochlorothiazide
Device: Amlodipine
  Arms: Amlodipine

SUMMARY:
The purpose of this study is to compare depressor effect and safety between combination therapy with telmisartan plus low-dose hydrochlorothiazide and amlodipine in hypertensive patients.

DETAILED DESCRIPTION:
In hypertensive patients whose blood pressure (BP) does not reach less than 140/90 mmHg with 5mg/day of amlodipine are divided the following two groups and BP response, laboratory data, and adverse effects are compared. Group 1: 12 week combination therapy with telmisartan plus low-dose hydrochlorothiazide. Group 2: Amlodipine is continuously administered.

ELIGIBILITY:
Inclusion Criteria:

* 5 mg/day of amlodipine is administered for more than 3 months
* Systolic or diastolic blood pressure >= 140/90 mmHg (more than 2 times measurements at outpatient clinic before start of the study)
* Outpatients

Exclusion Criteria:

* Secondary hypertension including renovascular hypertension with single kidney or bilateral stenosis
* Administration of antihypertensives other than amlodipine
* Cardiovascular disease (cerebral hemorrhage, cerebral infarction, TIA, angina, myocardial infarction, acute renal failure) occurs less than 6 months before start of the study
* Serum creatinine >= 2.0 mg/dl
* Severe hypertension (systolic or diastolic blood pressure >= 180/110 mmHg) or malignant hypertension (hypertensive organ damage is rapidly developing)
* Chronic heart failure (NYHA class>=III to VI)
* Contraindication of telmisartan or hydrochlorothiazide
* Hyper- (>= 5.5 mEq/L) or hypo- (<=3.5 mEq/l) potassemia
* Untreated hyperuricemia or uncontrolled hyperuricemia (serum uric acid >= 8.0 mg/dl)
* Diabetic patients who require insulin therapy, uncontrolled diabetic patients (hemoglobin A1c >=9.0%), or patients who possess the risk of hypoglycemic attack
* Patients inadequate for the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-07; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Changes in office blood pressure | After 12 week treatment

SECONDARY OUTCOMES:
1) Home blood pressure in early morning and before going to bed 2) Changes in uric acid, total cholesterol, HDL cholesterol, LDL cholesterol, triglyceride, fasting plasma glucose (only in diabetic patients), hemoglobin A1c (only in diabetic patients | After 12 week treatment

CONTACTS AND LOCATIONS:
Overall Officials: Toshiro Fujita, MD, PhD, Principal Investigator — Professor, Department of Nephrology and Endocrinology, University of Tokyo Graduate School of Medicine
Locations (1):
- Department of Nephrology and Endocrinology, University of Tokyo Graduate School of Medicine, Tokyo, Japan